CLINICAL TRIAL: NCT01246284
Title: Efficacy and Safety of Different Concentrations of Intralesional Triamcinolone Acetonide in Alopecia Areata: A Prospective, Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Efficacy and Safety of Different Concentrations of Localized Injections of Steroids in the Treatment of Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H10-02231
Record Dates: First submitted 2010-11-08; First posted 2010-11-23 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata; Intralesional; Triamcinolone acetonide; Concentration
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): Please note that the letter are assigned to different areas of injections within the same patient. All patients will be receiving the same treatment
  Interventions: Drug: Triamcinolone acetonide
- B (Active Comparator): Please note that the letter are assigned to different areas of injections within the same patient. All patients will be receiving the same treatment
  Interventions: Drug: Triamcinolone acetonide
- C (Active Comparator): Please note that the letter are assigned to different areas of injections within the same patient. All patients will be receiving the same treatment
  Interventions: Drug: Triamcinolone acetonide
- D (Placebo Comparator): Please note that the letter are assigned to different areas of injections within the same patient. All patients will be receiving the same treatment.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Triamcinolone acetonide — Injections will be given within a 3 cm2 area of alopecia which will be divided into 4 quadrants. Three different concentrations of triamcinolone acetonide will be used: 2.5, 5, and 10 mg/ml. Each quadrant will receive injections with either triamcinolone acetonide 2.5 mg/ml, triamcinolone acetonide 5 mg/ml, triamcinolone acetonide 10 mg/ml, or normal saline as a control. Injection of 0.1 ml will be given intradermally using a 30 gauge half inch long needle attached to a 3 ml syringe. Each quadrant will receive approximately 7 injections per treatment session so the total dose of triamcinolone acetonide will be around 13 mg. Injections will be given vertically, with the beveled side of the needle directed to the opposite side and 2 mm away from the margin of the adjacent quadrant to avoid a diffusion effect. The treatment will be repeated every 4 to 6 weeks for a total of 6 treatment sessions.
  Arms: A; B; C
Other: Normal saline
  Arms: D

SUMMARY:
Alopecia areata (AA) is a disease characterized by areas of hair loss. Localized steroid injections is the standard treatment for limited disease. There are no existing studies that compare different concentrations of steroids in the treatment of AA. This study will compare the efficacy and safety of different concentrations of localized steroid injections in the treatment of AA. Six treatment sessions will be done over 6 to 9 months. The investigators will compare the following concentrations: 2,5mg/ml, 5mg/ml, 10mg/ml, and normal saline.

DETAILED DESCRIPTION:
Alopecia areata (AA) is an autoimmune disease characterized by nonscarring hair loss with varying degree of severity. It most commonly involves scalp hair. It was estimated to occur in 0.1% to 0.2% of the general population in the united states. Patchy hair loss is the most common pattern seen in AA.

There are many treatment modalities available for AA, however, none of them cure the disease. Given the potential for spontaneous recovery in AA, studies assessing the efficacy of a certain therapeutic modality must be conducted in a controlled fashion. Treatment with intralesional corticosteroids (ILCSs) is considered the first-line therapy in adult patients with less than 50% scalp involvement. Use of ILCSs in AA was first reported by Kalkoff in 1958 using hydrocortisone. There are no published randomized controlled trials on the use of ILCSs in AA. Triamcinolone acetonide (TA) is the most commonly used form of ILCSs. It is characterized by low solubility, being slowly absorbed from the injection site, prompting maximal local action, limiting diffusion and spread through tissue, and not giving rise to systemic side effects if used in therapeutic doses. Use of intralesional (IL) TA in AA was first described by Orentreich et al. in 1960. IL TA is usually used in concentrations ranging from 2.5 to 10 mg/ml. Injections (0.1 ml per injection site) are given intradermally every 4 to 6 weeks. Abell and Munro used IL TA in the treatment of AA of varying degree of severity in 84 patients. The concentration used was 5 mg/ml and injections were given three times every 1 to 2 weeks. Fifteen patients received injections with isotonic normal saline as a control. Seventy one percent of patients with limited AA have shown evidence of regrowth compared to only 7% of patients in the control group. They also noticed that IL TA injections failed in all patients with rapidly progressive disease.

Side effects of IL TA include pain at the injection site, mild bleeding, transient atrophy and telangiectasia, hypopigmentation, hyperpigmentation. Infection is uncommon but caution over bony prominences is recommended. Adrenal suppression is rare when using lower doses. It has been reported in one patient who received a total dose of 22.5 mg in one session and the serum cortisol level normalized after 3 days. It has been shown that TA at a dose of 20 mg does not result in adrenal suppression. Hypersensitivity reactions to TA or the vehicle carboxymethylcellulose are extremely rare.

To our knowledge, there are no prospective studies comparing the efficacy and safety of different concentrations of IL TA in the treatment of AA. Helfman compared the therapeutic effect of different concentrations of IL TA in the treatment of different dermatoses. He included only one patient with localized AA. He injected TA using three different concentrations (2.5, 5, and 10 mg) and a diluent as placebo. Injections were done in 4 different quadrants within the same patch. He noticed that there was an equivalent degree of hair regrowth in the three sites injected with TA, and no regrowth in the site injected with the diluent.

Study Objectives

1. To compare the efficacy of different concentrations of IL TA in the treatment of AA.
2. To compare the side effect profile of different concentrations of IL TA when used in the treatment of AA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Less than 50% scalp involvement
* Patients should have a patch of at least 4.5 cm in the smallest diameter

Exclusion Criteria:

* Current episode of alopecia areata for longer than 2 years
* Evidence of hair regrowth at baseline
* Patients who received treatment with a topical, intralesional, or systemic agent within the past month
* Rapidly progressing disease
* Hypersensitivity to Triamcinolone acetonide or vehicle
* Pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Hair growth | 4-6 weeks after each treatment session

SECONDARY OUTCOMES:
Side effects | 4-6 weeks after each treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Shapiro, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Center, Vancouver General Hospital, 835 West 10th Ave, Vancouver, British Columbia, Canada